CLINICAL TRIAL: NCT03481400
Title: Provoked Migraine Attacks With Calcitonin Gene-related Peptide (CGRP) in Patients Who Have Tried Preventive Treatment With Anti-CGRP Monoclonal Antibodies.
Brief Title: CGRP-induced Migraine Attacks in Patients Who Have Tried Anti-CGRP Monoclonal Antibody Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Casper Emil Christensen, MD, PhD student, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: H-16014580
Record Dates: First submitted 2018-03-13; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Migraine
Keywords: Calcitonin gene-related peptide
MeSH Terms: conditions — Migraine Disorders | interventions — Calcitonin Gene-Related Peptide

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, crossover design.
Who Masked: Participant, Investigator
Masking Description: Double-blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcitonin gene-related peptide (Experimental): Calcitonin gene-related peptide infusion (1.5 micrograms/min for 20 mins)
  Interventions: Drug: Calcitonin Gene-Related Peptide
- Placebo (Experimental): Infusion with placebo (isotonic saline)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Calcitonin Gene-Related Peptide — Calcitonin gene-related peptide intravenous infusion (1.5 micrograms/min for 20 mins)
  Other Names: CGRP
  Arms: Calcitonin gene-related peptide
Other: Placebo — Isotonic saline
  Arms: Placebo

SUMMARY:
The investigators aim to investigate the incidence of migraine attacks after calcitonin gene-related peptide (CGRP) infusion in patients who have tried anti-CGRP monoclonal antibody treatment for the prevention of migraine.

DETAILED DESCRIPTION:
Calcitonin gene-related peptide (CGRP) plays a role in migraine pathophysiology. Infusions of CGRP can trigger migraine-like attacks in migraine patients and antibodies against CGRP or the CGRP receptor significantly reduces the number of migraine days per month when administered regularly. Some patients however, do not experience migraine attack after CGRP infusion, and some do not experience migraine reduction with antibodies. The underlying mechanisms of these effects are largely unknown.

The purpose of this study is to examine CGRP-induced migraine in patients who have evaluated the efficacy of anti-CGRP monoclonal antibody treatment for migraine using a purpose-developed standardized interview. The investigators will use a double-blind, placebo-controlled crossover study design to examine migraine susceptibility to CGRP in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine according to the international classification of headache disorders version 3-beta
* Subject has tried anti-CGRP antibodies for migraine
* Women of childbearing potential are on safe contraception

Exclusion Criteria:

* Women of childbearing potential who do not use contraception. Includes non-hysterectomized women who have not been menopausal for at least two years. Safe contraception includes condoms, intrauterine devices, p-pills, surgical sterilization or gestagen injections.
* Daily drug intake apart from contraceptives and preventive medication for migraine.
* Ingestion of any drug 4 half-lifes before study start apart from contraceptives.
* Pregnant or breast-feeding women
* Migraine on the study day or less than 48 hours before CGRP infusion.
* A history of cardiovascular and/or cerebrovascular disease
* Systolic blood pressure >150 mmHg and/or diastolic blood pressure > 100 mmHg on study day.
* Systolic blood pressure <90 mmHg and/or diastolic blood pressure < 50 mmHg on study day.
* A history of mental illness
* A history of any illness or condition that is deemed relevant for participation by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of migraine | From 0 to 12 hours after CGRP infusion
  Incidence of migraine after CGRP infusion
Area under the curve of headache intensity | From 0 to 90 minutes after infusion and from 90 minutes to 12 hours after infusion
  Area under the curve of headache intensity from 0-90 min and 90 min-12 hours post infusion

SECONDARY OUTCOMES:
Heart rate | From 0 to 90 minutes after infusion
  Heart rate (beats per minute)
Blood pressure | From 0 to 90 minutes after infusion
  Blood pressure (millimeter of mercury)

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, prof., Study Director — Danish Headache Center
Locations (1):
- Danish Headache Center, Rigshospitalet Glostrup, Copenhagen, Glostrup, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Christensen CE, Younis S, Deen M, Khan S, Ghanizada H, Ashina M. Migraine induction with calcitonin gene-related peptide in patients from erenumab trials. J Headache Pain. 2018 Nov 8;19(1):105. doi: 10.1186/s10194-018-0927-2. PMID 30409109